CLINICAL TRIAL: NCT05146414
Title: Clonal Hematopoiesis of Indeterminate Potential and Accelerated Atherosclerosis in Patients With Systemic Lupus Erythematosus
Brief Title: Clonal Hematopoiesis of Indeterminate Potential and Accelerated Atherosclerosis in Systemic Lupus Erythematosus
Acronym: HEMATOPLUS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Pr Nathalie COSTEDOAT-CHALUMEAU (Unknown)
Responsible Party: Sponsor
Other Study IDs: CRC18058
Record Dates: First submitted 2021-11-25; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; Clonal hematopoiesis of indeterminate potential; Cardiovascular events
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Accelerated atherosclerosis in patients with systemic lupus erythematosus (SLE) is not fully explained by Framingham risk factors. The detection in asymptomatic patients of somatic mutations in genes involved in hematopoietic malignancy- defining clonal hematopoiesis of indeterminate potential (CHIP) - predisposes to cardiovascular events (CVE) in general population. We aimed to determine whether CHIP is associated with CVE in SLE.

DETAILED DESCRIPTION:
SLE patients indeed display an accelerated atherosclerosis that strongly contributes to the excess mortality observed but is poorly explained by the traditional cardiovascular risk factors. Clonal hematopoiesis defines the clonal expansion of hematopoietic cells driven by a selective advantage given by leukemia-associated somatic mutations. Clonal hematopoiesis is said of indeterminate potential (CHIP) when found in asymptomatic patient. CHIP strongly correlated with age and logically predispose to haematological malignancy, but is also causally associated with cardiovascular events (CVE) in the general population. The main objective of our study was to determine whether CHIP is associated with CVE in SLE patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a systemic lupus erythematosus

Exclusion Criteria:

* Inadequate follow-up period (< 20 months) -past history of CVE at baseline for inclusion in the TROPOPLUS study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with a systemic lupus erythematosus
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2007-07-10 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the occurrence of cardiovascular events (CVE) over follow-up. | >20 months after PLUS inclusion
  Incidents CVE were ascertained by physician interview using a standardized questionnaire and through examination of medical records. CVE included coronary heart disease, stroke, revascularization procedure for other atherosclerotic cardiovascular diseases and sudden cardiac death. Coronary heart disease was defined as a history of angina, coronary revascularization, or myocardial infarction. All CVE that occurred through March 2019 were considered for analysis

SECONDARY OUTCOMES:
Prevalence of CHIP in SLE | at PLUS inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Karim SACRE, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat, Paris, France

REFERENCES:
- [Derived] David C, Duployez N, Eloy P, Belhadi D, Chezel J, Guern VL, Laouenan C, Fenwarth L, Rouzaud D, Mathian A, de Almeida Chaves S, Duhaut P, Fain O, Galicier L, Ghillani-Dalbin P, Kahn JE, Morel N, Perard L, Pha M, Sarrot-Reynauld F, Aumaitre O, Chasset F, Limal N, Desmurs-Clavel H, Ackermann F, Amoura Z, Papo T, Preudhomme C, Costedoat-Chalumeau N, Sacre K. Clonal haematopoiesis of indeterminate potential and cardiovascular events in systemic lupus erythematosus (HEMATOPLUS study). Rheumatology (Oxford). 2022 Nov 2;61(11):4355-4363. doi: 10.1093/rheumatology/keac108. PMID 35176141